CLINICAL TRIAL: NCT01850849
Title: A Phase I, First-in-Human, Vehicle Controlled, Single Ascending Dose Trial Evaluating the Safety, Tolerability and Pharmacokinetics in Male Subjects With AD and in Healthy Male Subjects of Cutaneous Application of LEO 39652 Cream
Brief Title: Safety, Tolerability and Pharmacokinetics in AD Subjects and Healthy Subjects of Cutaneous Application of LEO 39652 Cream
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: LEO Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: LP0083-1011
Record Dates: First submitted 2013-05-07; First posted 2013-05-10 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2015-01

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- LEO 39652 cream (Experimental): Active drug
  Interventions: Drug: LEO 39652 cream
- LEO 39652 cream vehicle (Placebo Comparator): Placebo drug
  Interventions: Drug: cream vehicle

INTERVENTIONS:
Drug: LEO 39652 cream
  Arms: LEO 39652 cream
Drug: cream vehicle
  Arms: LEO 39652 cream vehicle

SUMMARY:
The principle aim of this study is to obtain safety, tolerability and pharmacokinetic data when LEO 39652 cream is administered cutaneously as single dose to subjects with atopic dermatitis and to healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects or subjects with AD as defined by the Hanifen and Rajka criteria and with at least mild disease activity (IGA >2) for the whole body
* AD lesions amenable to cutaneous treatment located on the trunk and/or limbs (only for AD subjects)
* Male subjects aged between 18 and 65 years with a body mass index (BMI) between 19.0 and 32.0 kg/m2 inclusive

Exclusion Criteria:

* Subjects who currently suffer from, or show signs of eczema or other skin lesions (only for healthy subjects)
* Subjects who are still participating in a clinical trial (e.g. attending follow-up visits) or who have participated in a clinical study involving administration of an investigational product or a marketed drug product within the past 3 months prior to the first dosing occasion.
* Subjects with known immunocompromised state due to treatment with immunosuppressive drugs or due to history of a disease leading to immunocompromised status.
* History of or current cardiac arrhythmic disorder
* Subjects with a current active malignancy or a history of malignancy in remission for less than 5 years except excised skin (not melanoma) and cervical cancer.
* Subjects who have any clinically significant allergic disease (excluding non- active hayfever) as determined by the Investigator

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-05; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events and change from baseline in vital signs (blood pressure, pulse rate) ECG, clinical laboratory and local tolerability assessments | Up to 48 hours after dosing

SECONDARY OUTCOMES:
LEO 39652 and metabolites in blood | Up to 48 hours after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Chiesa, MD, Principal Investigator — Covance Clinical Research Unit, Hyde Street, Leeds, UK
Locations (2):
- United Kingdom (2):
  - Covance Clinical Research Unit, Hyde Street, Leeds, UK, Leeds
  - Covance Royal Liverpool Clinical Research Unit, Liverpool

IPD SHARING:
Plan to Share IPD: No